CLINICAL TRIAL: NCT02083432
Title: Cognitive Behavioural Treatment of Intra-oral Injection-phobia in 10-16 Year Old Children and Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bergen (Other)
Responsible Party: Principal Investigator, Marit Slåttelid Skeie, UBergen, University of Bergen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2010/63
Record Dates: First submitted 2014-02-25; First posted 2014-03-11 (Estimated); Last update posted 2018-08-16 (Actual); Status verified 2018-08

CONDITIONS: Dental Anxiety
Keywords: intra-oral injections; CBT; Blood-Injury-Injection-phobia; DSM-IV. 300.29

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 5-weeks waiting list control (Active Comparator): Half of the participants were randomly assigned to 5-weeks waiting list/Control group.The participants in the waiting list/Control Group are enrolled to the treatment Group (INtervention: 5 sessions of CBT) after 5 weeks if they still meet the diagnostic criteria of a specific phobia (according to DSM-IV).
  Interventions: Behavioral: 5 session of CBT performed by specially trained dentists
- 5 session of CBT (Experimental): Half of the participants were direct enrolled to 5 weeks(5 sessions) of cognitive behaviour therapy (CBT) performed by specially trained dentists. (Intervention: CBT)
  Interventions: Behavioral: 5 session of CBT performed by specially trained dentists

INTERVENTIONS:
Behavioral: 5 session of CBT performed by specially trained dentists — A total of 60 participants are randomly assigned to a 5-weeks waiting list Control Group or directly enrolled to the 5-session of CBT treatment Group.
  The participants in the waiting list Control Group are enrolled to the treatment Group (5 sessions of CBT) after 5 weeks if they still meet the diagnostic criteria of a specific phobia (according to DSM-IV).

SUMMARY:
The aims of the study: to explore the possible effectiveness of cognitive behavior treatment (CBT) among children and adolescents with formally diagnosed intra-oral injection phobia (DSM-IV), when performed by specially trained dentists.

The patients diagnosed with intra-oral injection phobia according to the diagnostic manual DSM-IV. The effect of cognitive behavior therapy when performed by specially trained dentists will be evaluated. Patients referred to the Centre for Odontophobia, and who meet the inclusion criteria, will be allocated to an immediate treatment group (test group) and a waiting list group (control group) of 30 subjects in each group. After treatment they will be followed up during a 1-year period.

Hypotheses are formulated based on the literature and previous population and treatment studies of similar designs among adults at the Centre for Odontophobia.

DETAILED DESCRIPTION:
The aims of the study: to explore the possible effectiveness of cognitive behavior treatment (CBT) among children and adolescents with formally diagnosed intra-oral injection phobia (DSM-IV), when performed by specially trained dentists.

The patients diagnosed with intra-oral injection phobia according to the diagnostic manual DSM-IV. The effect of cognitive behavior therapy when performed by specially trained dentists will be evaluated. Patients referred to the Centre for Odontophobia, and who meet the inclusion criteria, will be allocated to an immediate treatment group (test group) and a waiting list group (control group) of 30 subjects in each group. After treatment they will be followed up during a 1-year period.

Hypotheses are formulated based on the literature and previous population and treatment studies of similar designs among adults at the Centre for Odontophobia.

Inclusion criteria: referred 10-17-yr-olds (N=60) who refused intra-oral injections due to intra-oral injection-phobia. This randomized controlled study consisted of a test group (immediate treatment) and a control group (5 weeks waiting list). A diagnostic interview was performed by trained clinical psychologists, and 5 sessions of CBT were performed by 4 specially trained dentists. Each session had a maximum duration of one hour. Assessment at pre-treatment, post-treatment and 1-yr follow -up included responses from 4 different validated self-report instruments; Children's Fear Survey Schedule-Dental Subscale (CFSS-DS), Blood Phobia Scale (BS), Injection Phobia Scale for Children (IPS-C) and Intra-Oral Injection-Phobia Scale (IOIP). Paired sample t-tests were performed on the sumscores of the self-report instruments pre- , post waitlist, and post- treatment (n=17).

ELIGIBILITY:
Inclusion Criteria:

* Children between 10 and 16 years old diagnosed by clinical psychologist with Intra-oral injection phobia (DSM-IV 300.29).
* All patients refused to have intra-oral injections in Public Dental Health Clinics.
* Phobia of injections had to be the main phobia during dental treatment.

Exclusion Criteria:

* Accept anaesthetic infiltration during behavioural approach test.
* Cognitive impairment.
* Refuse to participate according to the study protocol.

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2013-12; Primary Completion 2016-06-30 (Actual); Study Completion 2016-06-30 (Actual)

PRIMARY OUTCOMES:
Intra-oral injection-phobia in children and adolescents. Prevalence, subgroups and the effect of cognitive behavioral treatment (CBT) | at 1 year follow-up
  Outcome measure: to evaluate whether children and adolescents diagnosed with intraoral injection phobia and treated with CBT, will be able to receive intraoral injections at an external dentist at 1 year follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Marit S Skeie, Professor, Principal Investigator — University of Bergen, Norway
Locations (1):
- University of Bergen, Bergen, Norway